CLINICAL TRIAL: NCT07165808
Title: Effect of Product Characteristics on the Abuse Liability of Nicotine Pouches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dae Hee Han, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009622; R00DA058241-03 (NIH); 2025P012303 (Other: Emory IRB)
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Nicotine Addiction
Keywords: Nicotine Addiction; Oral Nicotine Pouches; Behavioral Responses
MeSH Terms: conditions — Tobacco Use Disorder | interventions — pHLIP protein

STUDY DESIGN:
Intervention Model Description: Participants will take the intervention along two experimental factors: nicotine concentration (low [e.g., 3-4 mg] vs. high [e.g., 6-8 mg]) and pH level (low [<8.5] vs. high [≥8.5]). Each participant will be exposed to all four NP conditions in randomized order, with one condition administered per visit.
Masking Description: Participant and Investigator will remain blinded to the intervention dose and pH
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nicotine Pouches group (Experimental): Participants will self-administer NPs that differ along two experimental factors: nicotine concentration (low [e.g., 3-4 mg] vs. high [e.g., 6-8 mg]) and pH level (low [<8.5] vs. high [≥8.5]). Each participant will be exposed to all four NP conditions in randomized order, with one condition administered per visit.
  Interventions: Other: Nicotine pouch: Low dose; Other: Nicotine pouch: High dose; Other: Low pH; Other: High pH

INTERVENTIONS:
Other: Nicotine pouch: Low dose — Nicotine pouch: 3-4 mg
Other: Nicotine pouch: High dose — Nicotine pouch: 6-8 mg
Other: Low pH — Nicotine pouch with low pH level [<8.5]
Other: High pH — Nicotine pouch with high pH level [>8.5]

SUMMARY:
The goal of this study is to assess the effects of nicotine concentration and its interplay with pH on sensory experience, product appeal, and abuse liability of NPs among young adults NP users.

Primary objective is to assess the effect of variation in nicotine concentration in nicotine pouches (NPs) and its interaction effect with pH level on three proximal outcomes of relevance to regulation: (1) sensory experience, (2) product appeal, and (3) abuse liability of NPs.

DETAILED DESCRIPTION:
Oral nicotine pouches (NPs) are a rapidly growing segment of nicotine products regulated by the U.S. Food and Drug Administration (FDA). These microfiber pouches contain nicotine but no tobacco leaf, and they dissolve in the mouth without requiring spitting. Between late 2019 and early 2022, NP sales surged from 126 million to 808 million units. Their sleek packaging, concealability, and "tobacco-free" claims have made them particularly appealing to young adults, with recent studies showing that over 10% of young adults reported using NPs in the past 30 days. However, this popularity raises health concerns. NPs deliver nicotine efficiently through buccal absorption, leading to rapid increases in blood nicotine levels, which may contribute to oral toxicity, cardiovascular effects, and nicotine dependence. These factors also elevate the abuse liability of NPs-defined as the likelihood of non-medical use leading to harmful consequences.

The FDA has the authority to impose stricter regulations on products with characteristics that enhance appeal and sensory experience, especially among youth. For instance, the agency has proposed banning menthol cigarettes due to their ability to mask irritation and encourage deeper inhalation of nicotine. Similar regulatory scrutiny is now being applied to emerging products like NPs. One key factor influencing product appeal is nicotine formulation. Free-base nicotine, commonly used in non-combustible products like e-cigarettes (ECs), has aversive effects such as bitterness and airway irritation, especially at high concentrations. To counter this, manufacturers began adding organic acids to convert nicotine into a protonated salt, lowering the product's pH and improving its palatability. This shift not only enhances the sensory experience but also increases the abuse liability of high-nicotine products. Evidence suggests that regulating acid additives or setting minimum pH levels could reduce the appeal of these products. Since NPs also use acid additives to lower pH, they share similar characteristics with ECs that attract young users, underscoring the need for targeted regulatory action.

ELIGIBILITY:
Inclusion Criteria:

* Current established users of nicotine pouches (have used nicotine pouches in the past 30 days & currently use nicotine pouches every day or someday)
* Positive cotinine test via saliva test strip
* Those who are unmotivated to quit nicotine use
* Read and speak English.
* Poly-users of nicotine pouches, e-cigarettes (e.g., vape ≥20 days/month), and tobacco (e.g., ≥4 cigarettes/day for ≥2 years) will be eligible for participation

Exclusion Criteria

* Planning to cut down or quit using nicotine in the next 30 days
* Currently pregnant or breastfeeding
* History of stroke, seizures, high blood pressure, heart disease/problems, or cardiovascular disease contraindications for nicotine.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Abuse liability: Amount of time with Nicotine product | Visit 1, Visit 2, Visit 3, Visit 4 (all visits within 2-4 weeks)
  Total amount of time with Nicotine Pouches in mouth (excluding periods in between NPs after disposal)
Abuse liability: Number of Nicotine Pouches used | Visit 1, Visit 2, Visit 3, Visit 4 (all visits within 2-4 weeks)
  Total number of Nicotine Pouches used (i.e., larger number and longer time with Nicotine Pouches, higher abuse ability.
Subjective effects measures: Drug Effects Questionnaire | Visit 1, Visit 2, Visit 3, Visit 4 (all visits within 2-4 weeks)
  During the session, participants will also repeatedly (every 30 min) complete the subjective effects measures of abuse liability of NP (using VAS), which will be developed based on the Drug Effects Questionnaire (DEQ). A modified version of the DEQ will be used to rate acute responses to the NP on the Visual Analogue Scale (range, 0-100).
  Items assess liking/wanting (e.g., "I enjoy nicotine buzz," "I feel good effects from the NP," "I want more," "I feel the NP strength," and "I like the NP effect").
Subjective effects measures: Modified Cigarette Evaluation Questionnaire | Visit 1, Visit 2, Visit 3, Visit 4 (all visits within 2-4 weeks)
  Modified Cigarette Evaluation Questionnaire will also be used to measure domains of subjective reinforcing effects (product satisfaction, psychological reward; e.g., "NP is satisfying" on a 7-point scale (0-7).
Product appeal | Visit 1, Visit 2, Visit 3, Visit 4 (all visits within 2-4 weeks)
  After each administration, participants will use visual analogue scales (VAS, 0-100 range) to rate the product they just used: (1) "How much did you like the product?" (liking); (2) "How much did you dislike the product?" (disliking); and (3) "Would you use the product again?" (use again). A composite appeal score will also be calculated by averaging the 3 appeal ratings (Cronbach's α will be estimated to assess scale reliability; disliking will be reverse-scored).
Sensory Attribute | Visit 1, Visit 2, Visit 3, Visit 4 (all visits within 2-4 weeks)
  Participants will answer following sensory quality questions: (1) "How sweet was the product?"; (2) smooth?; (3) bitter?; and (4) harsh? (VAS 0-100, "Not at all" to "Extremely". Burning and tingling sensation will be measured at each trial.

SECONDARY OUTCOMES:
Nicotine product use history: Number of days | past 30-day
  Information will be collected on past 30-day number of days used nicotine pouches (NPs)
Nicotine product use history: Number of Nicotine product | past 30-day
  Number of Nicotine product used per day
Nicotine product use history: Amount of time with Nicotine product | past 30-day
  Amount of time with Nicotine product in mouth per episode
Nicotine Pouches brand | past 30-day
  Data on brand names of NPs will be collected
Number of e- cigarettes | past 30-day
  Number of e- cigarettes used in past 30 days.
Tobacco use | past 30-day
  Number of tobacco products used in last 30 days

OTHER OUTCOMES:
Salivary cotinine | Baseline
  Test strips that provide a semiquantitative index of salivary cotinine will be collected to provide descriptive data on nicotine exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Han, PhD, Principal Investigator — Rollins School of Public Health
Locations (1):
- Rollins School of Public Health, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level data collected as part of the R00 study, including baseline demographics, behavioral measures, and experimental outcome variables.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available within 12 months after publication of the primary study results and will remain available for at least 3 years thereafter.
Access Criteria: Data will be shared through a secure, controlled-access repository. Researchers must submit a data use request, obtain approval from the principal investigator, and sign a data use agreement to ensure protection of participant confidentiality and compliance with IRB and NIH policies